CLINICAL TRIAL: NCT04790461
Title: The Effect of an Application Based on Training and Progressive Relaxation Exercises on the Quality of Life, Perceived Stress and Coping Ways of Caregivers of Mentally Handicapped Individuals: A Randomized Controlled Study
Brief Title: The Quality of Life, Perceived Stress and Coping Ways of Caregivers of Mentally Handicapped Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafkas University (Other)
Collaborators: Sakarya University (Other)
Responsible Party: Principal Investigator, Gönül GÖKÇAY, Lecturer, Kafkas University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: 80576354-050-99/254
Record Dates: First submitted 2021-03-06; First posted 2021-03-10 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Intellectual Disability
Keywords: caregivers; model-based education; progressive relaxation exercises; quality of life; stress; mobile health; Intellectual Disability
MeSH Terms: conditions — Intellectual Disability | interventions — Evaluation Studies as Topic

STUDY DESIGN:
Intervention Model Description: 1. experimental group: face-to-face training + PMR exercise
  2. experimental group: mobile health education + PMR exercise
  3. experimental group: face-to-face and mobile health training + PMR exercise control group
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants were assigned to groups using the "simple randomization method". Participants were not informed of which group they were in. Automated computer-based randomization resulted in the implementation of the experiment with the scheduling scenario and confidential allocation of participants to one of the four intervention branches. The researcher was blind to all conditions until the participants started the computer program and the intervention began. Participants were also unaware of whether the group they were assigned to was an experimental or a control condition. In addition, researchers coding and analyzing data will be blind to randomization and interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 1. experimental group: face to face education+PMR exercise (Experimental): The education and PMR exercises prepared in line with the face-to-face Roy adaptation model will be applied. In groups of 8-10 people, the first 4 sessions in rehabilitation centers will last for the first 4 sessions, and then PMR exercises will be taught and applied (between the 2nd and the 5th weeks, they will be encouraged to do PGE twice at home). The next 4 weeks will be provided with PMR consultancy (3 times a week application / total 24 sessions of PMR application). PMR exercises will be given a follow-up schedule and the caregivers will be followed up by the caregivers themselves and the researchers.
  Interventions: Other: Pre-post test; Behavioral: face-to-face training + PMR exercise
- 2. experimental group: mobile health education + PMR exercise (Experimental): Access to mobile applications will be provided for 8 weeks, including the Roy adaptation model-based training and PMR exercises, which include video and training presentations prepared by the consultant and researcher, as a power point presentation. PMR exercises will be uploaded to the system by uploading a follow-up schedule to the system, and it will be ensured that the person can follow himself / herself at least 3 times a week (24 sessions in total) and the researchers can follow the participants.
  Interventions: Other: Pre-post test; Behavioral: mobile health education + PMR exercise
- 3rd experimental group: face to face and mobile health education + PMR exercise (Experimental): 4 sessions prepared in line with the Roy adaptation model face to face and held in rehabilitation centers, training in groups of 8-10 people, teaching PMR exercises and installing phone applications that can be accessed for 8 weeks), 8-week intervention including training (enabling them to do progressive relaxation exercises and access to training content) will be provided. . The PMR exercises will be uploaded to the system / given as a printout according to the caregiver's preference, and it will be ensured that the person can follow himself / herself at least 3 times a week (24 sessions in total) and the researchers watch the participant.
  Interventions: Other: Pre-post test; Behavioral: face-to-face and mobile health education + PMR exercise
- Control group (Other): Without applying any intervention, the post-test YBYKA, ASÖ and SBÇYA scales will be applied in the 10th week of the study. After all the tests for the study are measured and finished, they will be provided with training and relaxation exercises.
  Interventions: Other: Pre-post test

INTERVENTIONS:
Other: Pre-post test — Adult Caregiver Quality of Life Questionnaire (AC-QoL) Perceived Stress Scale (PSS) The Stress Coping Styles Questionnaire (SCSQ)
Behavioral: face-to-face training + PMR exercise — 4 weeks Roy adaptation-based face-to-face training + PMR exercises to be taught, 4 weeks exercise counseling
  Arms: 1. experimental group: face to face education+PMR exercise
Behavioral: mobile health education + PMR exercise — To provide awareness and exercise with 8 weeks Roy adaptation model-based training and mobile application access with PMR exercise content
  Arms: 2. experimental group: mobile health education + PMR exercise
Behavioral: face-to-face and mobile health education + PMR exercise — 4 weeks face-to-face training based on Roy adaptation model + teaching PMR exercises and 4 weeks based training on Roy adaptation model and mobile application access with PMR exercise content
  Arms: 3rd experimental group: face to face and mobile health education + PMR exercise

SUMMARY:
Disability is a dynamic, multidimensional and diverse public health problem. Although the primary care burden of the disabled is mostly on mothers, caregivers cannot find little or no support socially and they have a high risk of experiencing physical and psychological health problems. In the studies carried out; Disabled caregivers reported higher and lower quality of life than healthy individuals' relatives with physical ailments such as asthma, arthritis, back pain, care burden, pain, insomnia, fatigue, depression, anxiety, stress. This study was planned to determine the effect of an application based on research, education and progressive relaxation exercises on the quality of life, perceived stress and coping strategies of caregivers of mentally disabled individuals.

HYPOTHESES OF THE RESEARCH H1:Face to face education and PGE exercises applied to mentally disabled individual caregivers have an effect on caregivers' quality of life, perceived stress and ways of coping with stress.

H2:Mobile application applied to mentally disabled caregivers and Education and PGE exercises have an effect on the quality of life of caregivers, their perceived stress and ways of coping with stress.

H3:The Face to face + Mobile Application education and PGE exercises applied to mentally disabled individual caregivers have an effect on the caregivers' quality of life, their perceived stress and ways of coping with stress.

DETAILED DESCRIPTION:
Disability, a dynamic, multidimensional and diverse public health problem, can be acquired temporarily/chronicly or later in life due to congenital, acute illness and/or injury. Although the primary care burden of the disabled is mostly on mothers, caregivers cannot find little or no support socially and they have a high risk of experiencing physical and psychological health problems. In the studies carried out; Disabled caregivers reported higher and lower quality of life than healthy individuals' relatives with physical ailments such as asthma, arthritis, back pain, care burden, pain, insomnia, fatigue, depression, anxiety, stress. It was determined that 64.3% of mentally disabled caregivers experience severe stress. The measure that improves family caregivers' knowledge about effective and safe care strategies can reduce/prevent stress-related problems and improve their quality of life. Roy's Adaptation model (RAM) is one of the most widely used nursing models to cope with various diseases and problems, which is applied to improve the quality of life and reduce stress in caregivers. Progressive relaxation exercise (PGE), which is an excellent step to cope with stress and stress, has been recognized as an effective technique used in controlling muscle tension. Stress (Novais et al., 2016; Wicaturatmashudi&Erman,2020; Özgündoğdu&Metin, 2019; Fernández Sánchez et al., 2020) and quality of life (Ghezeljeh et al., 2017; Bahrami-Eyvanekey et al., 2017). As a part of the holistic care of children with mental disabilities, the needs and problems of their primary caregivers should be taken into consideration and solutions should be developed. At the end of this study, the effectiveness of structured interventions consisting of different learning styles (face-to-face, mobile application, face-to-face and mobile application; education + PGE exercises) and relaxing exercises that alleviate the physiological and psychological burden of care were tested, and it was the most effective in increasing the quality of life and reducing stress of caregivers of mentally disabled individuals. method will be determined. The method that has been proven to be effective will be supported by mobile application for the widespread access of mentally disabled individuals to their caregivers, to reach more target groups.

In this study, randomized controlled, 3 experimental, 1 control group, pretest-posttest experimental design will be used as research design. The study will be conducted with the caregivers of mentally disabled individuals rehabilitated in rehabilitation centers. The sample size was calculated as 34 individuals in each group (136 individuals) with the G-Power 3.1.9.2 power analysis program. The data will be obtained using the personal information form, adult caregiver quality of life questionnaire, perceived stress scale, ways of coping with stress questionnaire. The data will be evaluated using SPSS statistics 20 program and Statistical significance will be accepted as p<.05.

ELIGIBILITY:
Inclusion Criteria:

* Having a child receiving education in a rehabilitation center in the province of Kars,
* Being a caregiver between the ages of 18-65,
* The individual he cared for should not have any disability other than mental disability
* Volunteering to participate in research,
* To be literate, to follow mobile application instructions,
* To have the knowledge to use the mobile application independently or to have another individual in the family who can help in this regard

Exclusion Criteria:

* Having a disability other than mental disability of the individual he cared for,
* Individuals with cognitive and physical dysfunction that will prevent interview or test application,
* Not wanting to participate in research.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2020-11-25 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Adult Caregiver Quality of Life Questionnaire (AC-QoL) | ten weeks
  Developed by Stephen Joseph et al. (2012), validity and reliability in Turkish by Gençer and Şengül, caregiver quality of life in 8 different areas (care giving, caring preference, patient care stress, financial issues, personal development, valuing, caregiving ability and caregiver satisfaction) is a questionnaire that provides the opportunity to evaluate. In scale evaluation, 0-40 points indicate "low quality of life", 41-80 points "average quality of life" and 81-120 points indicate "high quality of life" (Joseph et al. 2012; Gençer, 2020).
Perceived Stress Scale (PSS) | ten weeks
  Scale developed by Cohen, Kamarcık and Mermelstein (Cohen at al., 1983). A total of 14 items were designed to measure how stressful certain situations in a person's life are perceived. PSS scores are between 0 and 56. A high score indicates a person's high perception of stress (Eskin et al., 2013). In the original form of the scale, the internal consistency Cronbach alpha coefficient was 0.84, and the test-retest reliability coefficient was determined as 0.85 as a result of two measurements performed two days apart (Cohen at al., 1983). Cronbach coefficient alpha was found 0.87 (Eskin et al., 2013) and 0.722 (Yımaz 2020) in the Turkish validity and reliability study.
The Questionnaire of Ways to Cope with Stress (SBÇYA) | ten weeks
  The Coping Ways Questionnaire (WCQ) developed by Folkman and Lazarus was adapted into Turkish by Şahin and Durak (1995). The scale consists of five sub-dimensions: "confident", "optimistic", "helpless", "obedient" and "seeking social support". In the 30-item scale, the answers given for each item are in four-order evaluation (0- 30-70-100%) ranging from 0 to 100%.

CONTACTS AND LOCATIONS:
Overall Officials: Gönül GÖKÇAY, Principal Investigator — Kafkas University-Ataturk Health Services Vocational School Kars, Turkey, 36500; Ayşe ÇEVİRME, Study Director — Sakarya University Health Faculty of Health Science Sakarya, Turkey, 54100
Locations (2):
- Turkey (Türkiye) (2):
  - Kafkas University-Ataturk Health Services Vocational School, Kars, Turkey/Kars
  - Sakarya University Health Faculty of Health Sciences, Sakarya

IPD SHARING:
Plan to Share IPD: No
This protocol study is a doctoral thesis. Therefore, the process may take longer and there may be plagiarism at the article stage. Only the name of the study can be shared with other researchers. Please let's hide the rest of the protocol publication, I wish you the best of luck.

REFERENCES:
- [Background] Novais PG, Batista Kde M, Grazziano Eda S, Amorim MH. The effects of progressive muscular relaxation as a nursing procedure used for those who suffer from stress due to multiple sclerosis. Rev Lat Am Enfermagem. 2016 Sep 1;24:e2789. doi: 10.1590/1518-8345.1257.2789. PMID 27598379
- [Background] Ozgundondu B, Gok Metin Z. Effects of progressive muscle relaxation combined with music on stress, fatigue, and coping styles among intensive care nurses. Intensive Crit Care Nurs. 2019 Oct;54:54-63. doi: 10.1016/j.iccn.2019.07.007. Epub 2019 Jul 29. PMID 31371164
- [Background] Fernandez Sanchez H, Hernandez CBE, Sidani S, Osorio CH, Contreras EC, Mendoza JS. Dance Intervention for Mexican Family Caregivers of Children With Developmental Disability: A Pilot Study. J Transcult Nurs. 2020 Jan;31(1):38-44. doi: 10.1177/1043659619838027. Epub 2019 Apr 4. PMID 30947622
- [Background] Najafi Ghezeljeh T, Kohandany M, Oskouei FH, Malek M. The effect of progressive muscle relaxation on glycated hemoglobin and health-related quality of life in patients with type 2 diabetes mellitus. Appl Nurs Res. 2017 Feb;33:142-148. doi: 10.1016/j.apnr.2016.11.008. Epub 2016 Nov 14. PMID 28096008
- [Background] Bahrami-Eyvanekey Z, Ramezani-Badr F, Amini K, Karimian E. Comparison of the Effects of Guided Imagery and Progressive Muscle Relaxation on Quality of Life of Patients Undergoing the Coronary Artery Bypass Graft Surgery: A Randomized Clinical Trial. Iranian Journal of Nursing Research.2017; 12(3): 7-15.